CLINICAL TRIAL: NCT06886087
Title: Prospective Study to Assess the Risks of Perinephric Fat Thickness on Adverse Renal Outcomes Post Donor Nephrectomy - ProActive Study
Brief Title: Assessment of Risks of Perinephric Fat Thickness to Adverse Renal Outcomes Post Donor Nephrectomy
Acronym: ProActive
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aleksandra Kukla, Consultant Nephrology, Mayo Clinic
Other Study IDs: 24-006635
Record Dates: First submitted 2025-02-05; First posted 2025-03-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Living Kidney Donation; Hypertension; Nephrectomy
Keywords: healthy volunteers; kidney donation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, fat and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Obese: Participants with a BMI under 30
- Obese: Participants with a BMI greater than or equal to 30

SUMMARY:
The goal of this observational study is to learn if PRAT thickness is a marker of visceral obesity and its influence on donors' kidney function and blood pressure in living kidney donors. Population includes male/female, 18 years and up, living kidney donors scheduled for nephrectomy within 6 months. The main area it aims to help in, is future care managing blood pressure and obesity in living kidney transplant donors.

Primary Hypothesis: We hypothesize that Perirenal Fat Thickness (PRAT) may exhibit expansion, remodeling and inflammation that can negatively affect renal outcomes in LKDs.

Researchers will compare PRAT morphology and inflammation in LKDs with low and high PRAT thickness.

We will also correlate PRAT thickness with renal outcomes including vascular remodeling, at the time of donation and worsening hypertension and inadequately increased compensatory GFR of the LKD at 4-6 months post-donation.

Participants will be separated into one of two groups depending on their PRAT measurement and asked to give samples of their blood, perinephric fat, and urine as research samples. Clinically we will abstract data up to 12 months prior and 6 months after their nephrectomy that includes laboratory findings, CT measurements, vitals, exam data, demographics, medical history and current medications.

DETAILED DESCRIPTION:
6.1 Screening Visit Patients who have had their donor nephrectomy scheduled will be approached for enrollment. Potential participants must preliminarily meet all inclusion and no exclusion criteria to be approached by a study team member about study participation. If there is 10% (or greater) weight loss between the clinical donor evaluation visit and the potential screening visit the individual will not be approached for enrollment.

If all required inclusion and no exclusion criterion are met, the study team will present the consent form to the potential participant.

After the consent form has been signed, the following study procedures will be performed at the screening visit:

* The following information will be collected study team member will review the participant's demographic information, m The following information will be recorded from the participant's from their electronic medical record

  * Participant's demographic information
  * Medical history and current medications and, if needed, ask the participant clarifying questions
  * Pregnancy test results (if applicable)
  * Current medications
  * Most recent weight
  * Height
  * BMI
  * Clinical Donor Evaluation
  * PRAT Measurement
* The following lab results will also be collected from the medical record

  * Creatinine with eGFR
  * Comprehensive Metabolic Panel Glucose
  * Fasting Lipid Profile
  * HbA1c
  * 24-hour Urine for Albumin Excretion
* An 18-hour ABPM may be completed with subject consent at either the Screening Visit or Visit 1 if (if it has not been obtained clinically 6 months prior to the scheduled donor nephrectomy) or there has been a clinically significant blood pressure medication changes. A sphygmomanometry measurement will be collected at each visit unless the 18-hour ABPM is performed.

Serious adverse events will also be recorded and addressed as applicable at every study visit after the participant signs consent. All adverse events will be recorded from Visit 2 until the subject completes or is withdrawn from the study.

In applicable situations (i.e., the subject does not need to be seen in person to complete all study procedures) the screening visit can be completed remotely.

After this information has been collected, participants will be categorized into 1 of the 2 groups based upon their PRAT measurement and BMI. If the PRAT thickness or the BMI does not meet study criterion, the participant will be considered a screen failure.

6.2 Visit 1

During this visit, the following study procedures will also occur:

* The study team will record the following information from the medical record:

  * Changes in the participant's medical history or medications.
  * Participant's current weight and height.
  * Participant's BMI
* 10 mL of blood and 50mL urine will also be collected for research purposes.
* An optional 18-hour ABPM may be completed if the subject has consented to this procedure and it was not collected during the screening visit. If a subject declines the 18-hour ABPM a sphygmomanometry measurement will be collected.

6.3 Visit 2

Visit 2 will occur the day of the living kidney donor's nephrectomy. During this visit, the study team will perform the following:

* Record the following information from the participant's medical record:

  * changes to the medical history or medications.
  * The participant's current weight and height
  * Participant's BMI
  * Information on the nephrectomy.
  * Hemoglobin
  * 24-hour ABPM
* During the nephrectomy, the study team will collect a 5-10g fat sample for research analysis.

6.5 Visit 3

This visit will take place approximately 6 months after the donor nephrectomy. During this visit, the study team will:

* Record the following information from the EMR:

  * Any changes to the participant's medical history or medications.
  * The participant's current weight and, height.
  * Current BMI
  * The participant's blood pressure, via sphygmomanometry.
  * Creatinine with eGFR
  * Fasting Lipid Profile
  * Glucose
* An 18-hour APBM will be completed with participant consent and if it was not completed as a part of clinical care. If a subject declines the 18-hour ABPM a 6h AMBP monitoring performed clinically will be collected
* 10 mL of blood and 50 mL of urine will be collected for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will be restricted to living kidney transplant donors (LKDs). .

Exclusion Criteria:

* Those who do not meet Mayo Clinic Rochester's clinical criterion for donor nephrectomy.
* >10% weight change between the donor evaluation and donor nephrectomy
* Individuals who are pregnant or are planning to become pregnant
* Inability to comply with study procedures or any condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Living kidney donors scheduled for nephrectomy ages 18 - 80
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Proinflammatory Macrophage infiltrations of Perinephric Fat for LKD | 12 months
  Compare LKD total PRAT thickness with incidence of increased macrophages

SECONDARY OUTCOMES:
Development of new or worsening hypertension in LKD | 12 months
  Compare LKD total PRAT thickness with incidence of new or worsening HTN

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Kukla, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benavides X, Rogers RT, Tan EK, Merzkani MA, Thirunavukkarasu S, Yigitbilek F, Smith BH, Rule AD, Kukla A, Chow GK, Heimbach JK, Taner T, Dean PG, Prieto M, Stegall MD. Complications After Hand-Assisted Laparoscopic Living Donor Nephrectomy. Mayo Clin Proc. 2022 May;97(5):894-904. doi: 10.1016/j.mayocp.2021.11.023. Epub 2022 Apr 25. PMID 35483987
- [Background] Taler SJ, Messersmith EE, Leichtman AB, Gillespie BW, Kew CE, Stegall MD, Merion RM, Matas AJ, Ibrahim HN; RELIVE Study Group. Demographic, metabolic, and blood pressure characteristics of living kidney donors spanning five decades. Am J Transplant. 2013 Feb;13(2):390-8. doi: 10.1111/j.1600-6143.2012.04321.x. Epub 2012 Nov 8. PMID 23137211
- [Background] Ibrahim HN, Foley RN, Reule SA, Spong R, Kukla A, Issa N, Berglund DM, Sieger GK, Matas AJ. Renal Function Profile in White Kidney Donors: The First 4 Decades. J Am Soc Nephrol. 2016 Sep;27(9):2885-93. doi: 10.1681/ASN.2015091018. Epub 2016 Feb 17. PMID 26888476
- [Background] Locke JE, Reed RD, Massie AB, MacLennan PA, Sawinski D, Kumar V, Snyder JJ, Carter AJ, Shelton BA, Mustian MN, Lewis CE, Segev DL. Obesity and long-term mortality risk among living kidney donors. Surgery. 2019 Aug;166(2):205-208. doi: 10.1016/j.surg.2019.03.016. Epub 2019 May 7. PMID 31072668
- [Background] Sanchez OA, Ferrara LK, Rein S, Berglund D, Matas AJ, Ibrahim HN. Hypertension after kidney donation: Incidence, predictors, and correlates. Am J Transplant. 2018 Oct;18(10):2534-2543. doi: 10.1111/ajt.14713. Epub 2018 Apr 6. PMID 29498216
- [Background] Issa N, Sanchez OA, Kukla A, Riad SM, Berglund DM, Ibrahim HN, Matas AJ. Weight gain after kidney donation: Association with increased risks of type 2 diabetes and hypertension. Clin Transplant. 2018 Sep;32(9):e13360. doi: 10.1111/ctr.13360. Epub 2018 Aug 18. PMID 30053320
- [Background] Punjala SR, Adamjee Q, Silas L, Gokmen R, Karydis N. Weight trends in living kidney donors suggest predonation counselling alone lacks a sustainable effect on weight loss: a single centre cohort study. Transpl Int. 2021 Mar;34(3):514-524. doi: 10.1111/tri.13816. Epub 2021 Feb 3. PMID 33423338
- [Background] Liu BX, Sun W, Kong XQ. Perirenal Fat: A Unique Fat Pad and Potential Target for Cardiovascular Disease. Angiology. 2019 Aug;70(7):584-593. doi: 10.1177/0003319718799967. Epub 2018 Oct 9. PMID 30301366
- [Background] Ma S, Zhu XY, Eirin A, Woollard JR, Jordan KL, Tang H, Lerman A, Lerman LO. Perirenal Fat Promotes Renal Arterial Endothelial Dysfunction in Obese Swine through Tumor Necrosis Factor-alpha. J Urol. 2016 Apr;195(4 Pt 1):1152-9. doi: 10.1016/j.juro.2015.08.105. Epub 2015 Sep 28. PMID 26417644
- [Background] Wang D, Iversen J, Wilcox CS, Strandgaard S. Endothelial dysfunction and reduced nitric oxide in resistance arteries in autosomal-dominant polycystic kidney disease. Kidney Int. 2003 Oct;64(4):1381-8. doi: 10.1046/j.1523-1755.2003.00236.x. PMID 12969157